IRB CODE NUMBER: 2019.053

NCT number: 05530603

University of South Dakota Department of Social Work

Intervention To Promote Breast Cancer Screening Among American Indian Women

Study Protocol

Date of Document: 05/02/2022



| Office Use Or | ıly |
|---------------|-----|
| Date Received | l: |
| Protocol Num | ber |

# **Non-Medical IRB Submission Form**

Submit one copy of the application and required materials to <a href="https://example.com/humansubjects@usd.edu">humansubjects@usd.edu</a>. The signature page may be emailed or delivered to Slagle 107. <a href="https://example.com/studies not will be approved until we have received the signature page">https://example.com/studies not will be approved until we have received the signature page.</a>

| Today's Date: | | | | | |
|---|---|---|---|---|---|
| 08/7/2019 | | | | | |
| Project Title: | | | | | |
| | | | Among American Indian | | |
| Note: A student's ac | visor is cons | idered the "Princi | pal Investigator" and ha | s ultimate responsibility for the o | conduct of the student(s). |
| Principal Investiga<br>Department: Social<br>Qualifications to do<br>CITI Date: 10 May 2 | <b>Nork</b> email:<br>ne research: | Soonhee.Roh@<br>Principal | Investigator | 5-357-1593<br>date. (2 years for VA employe | es) |
| Other Investigator:<br>Department: | email: | | phone: | Role in Study: | CITI Date: |
| Other Investigator:<br>Department: | email: | | phone: | Role in Study: | CITI Date: |
| Other Investigator:<br>Department: | email: | 1981783 | phone: | Role in Study: | CITI Date: |
| Other Investigator:<br>Department: | email: | | phone: | Role in Study: | CITI Date: |
| FOR VA STUDIES | | | | | |
| | ease attach a | a copy of their ap | d Privacy Officer?<br>proval with signature pa<br>RB until approval has b | _ | |
| Section 1: General | Questions | | | | |
| | • | | | erest associated with this study<br>osure of Financial Interests) | ? |
| <ul> <li>Is this study externally funded? (If yes, please attach a copy for each one selected)</li> <li>□ No</li> <li>☑ Federally Sponsored Project-pending</li> <li>□ Industry Sponsored Study</li> <li>□ State Sponsored Project</li> </ul> | | | | | |
| committee | ?<br>N/A | | e their thesis or dissertat Yes lication until approval | tion, has it been approved by th | e dissertation or thesis |



| Office Use Only |
|-----------------|
| Date Received: |
| Protocol Number |

| 4. | . Have you, or do you, plan to submit this s<br>⊠ Yes – please submit a copy o<br>□ No | and the second s | oved consent/assent. |
|---|---|---|---|
| 5. | | eb App Breast Cancer | dy are to develop and evaluate the feasibility<br>Screening (wMammogram) intervention that |
| 6. | task(s) they will be expected to perform. (addresses two specific aims with a multi-meth period. The two phases are: (1) developing the wMammogram (Aim 2). Phase 1 incorporates with various stakeholders in Al communities the randomized clinical trial (RCT) design with Al (IRB), Dr. Roh will convene two focus groups and local health professionals with backgroun firsthand information about the general public as well as barriers, motivators, and possible to | (How will you contact them? nod, two-phase research project whammogram intervention is a Community Based Participa o design a culturally informed a women. In phase one, after the (N=20; n=10 for each group), lads in cancer and health manage the latter of | last contact with participant(s) please describe the What will you have them do?) The proposed study of that will take place in South Dakota over a three-year (Aim 1) and (2) evaluating the feasibility and efficacy of the story Research (CBPR) approach and a series of focus groups and practically refined intervention. Phase 2 uses a e approval of the Yankton Tribal Institutional Review Board Each group will consist of Al community leaders/members gement. The purpose of the two focus groups will be to obtain efs, attitudes, and values about breast cancer and screening, two, the wMammogram intervention will be implemented with the a mixed methods approach will be conducted at three and post-intervention focus group. |
| 7. | Have you attached letters of approval from ☐ Yes | m any schools or businesse<br>⊠ N/A | s involved? |
| Section | 2: Participants | 8 | |
| 8. | Please state the maximum number of par | ticipants you plan on enrolli | ng. <b>107</b> |
| 9. | Please describe the study populations by ☐ Males ☐ Non-English Speaking | checking all that apply. ⊠ Females □ Students in Grades K | ☐ University Students<br>-12 |
| 10 | D. Are you <b>specifically</b> targeting an ethnic g ☑ American Indian ☐ Alaskan Native ☐ Hispanic | group? Check any that apply ☐ African American ☐ Asian ☐ Other | /. □ Caucasian □ Pacific Islander |
| 11 | <ul> <li>1. Age ranges of subjects to be enrolled?</li> <li>☐ Birth-3</li> <li>☐ Middle School 10-13</li> <li>☑ Senior Citizens 64 and up</li> </ul> | <ul><li>□ Preschool 3-5</li><li>□ High School 14-17</li></ul> | ☐ Elementary 5-10<br>☑ Adult 18 and 64 |
| 12 | past two years, (4) who live in South Dakota,<br>own mobile phone or a mobile phone borrows<br>40-70 was selected based on the breast cano | omen, (2) who are aged 40 to (5) who are willing to possess ed from the research team for the er screening guidelines of the exclusion criteria include those | 70 years, (3) who have not received a mammogram in the an active email account, and (6) who are willing to use their he wMammogram intervention. The participant age range of American Cancer Society (ACS) that recommend women to se who (1) are minors (under 18 years), (2) received a |
| 13 | 3. Are any of the vulnerable populations liste | ed below going to be enrolle | ed in this study? |



| Office Use Only |
|-----------------|
| Date Received: |
| Protocol Number |

| | <ul> <li>☐ Your employees</li> <li>☐ Your students</li> <li>☐ Pregnant women</li> <li>☐ Prisoners</li> <li>☐ Children</li> <li>☐ Individuals with diminished mental/physical capacity</li> <li>☐ Pregnant women</li> <li>☐ Economically/educationally disadvantaged persons</li> </ul> |
|---|---|
| 14. | Are the research participants your students or employees? ☑ No ☐ Yes – explain how you plan on avoiding your student(s) feeling or perceiving undue influence for participation |
| 15. | Where will the research take place? Yankton Sioux Tribe |
| 16. | If this research is taking place in a classroom, describe what non-participants will do during the research (activities and supervisions). Students not participating in the research should not be singled out or penalized. N/A |
| 17. | Will the participant(s) receive any compensation or extra credit? If so please describe what type (i.e. SONA extra credit, gift card, monetary). If you are offering extra credit, please describe the non-research alternative way to earn the extra points. Please be sure to state this in the consent form along with a statement that students may stop participating at any time without losing the extra credit. To encourage participation, participants will be offered \$20 cash as an honorarium at three intervals (total \$60): baseline, one-week post-intervention, six-month follow-up survey, and \$50 for initial development of web mammogram focus group and post-intervention focus group. |
| Section 3 | Recruitment |
| 18. | How do you have access to the study population? In collaboration with the Community Advisory Board, participants will be recruited through flyers, newspapers, radio announcements, social service agencies, ethnic community organizations, colleges, and ethnic events. Flyers and announcements will describe the purpose of the project, eligibility criteria, and contact information. Interested Al women will call the telephone number provided, and recruitment staff will screen potential participants over the phone to determine whether they meet the inclusion criteria. |
| 19. | Are you obtaining subjects from private records (i.e. through your job, volunteer work, internship, etc.)? The data could be consider private records unless it is publicly available to anyone. □ Yes: Describe how you have permissible access. □ No |
| 20. | How will you initially contact and select the participants? (i.e. letter, e-mail, or advertisement). You must include all recruitment, announcements, and invites with your IRB application. Make sure they include the word "research", your study purpose, estimated time commitment, eligibility criteria, and your contact information for questions Participants will be recruited through flyers, newspapers, radio announcements, social service agencies, ethnic community organizations, colleges, and ethnic events. Flyers and announcements will describe the purpose of the project, eligibility criteria, and contact information. Interested Al women will call the telephone number provided, and recruitment staff will screen potential participants over the phone to determine whether they meet the inclusion criteria. |
| 21. | Describe how the subject's privacy will be protected? (I.e. testing or interviewing in private) <i>Privacy is about the person NOT the datathink about where the procedures will be conducted.</i> Participants will conduct a survey in a private conference. |
| 22. | Will there be a link to identify subjects? This could be a name, code, or reference that might be used to identify the subject outside of the context of the research setting. The key question is, "Is there any way that anyone, including the investigator, could start with a data record and trace it back to the person being studied?" If yes, then there is an identifier linked to the subject. |
| 1 | ☐ Yes: Explain the link and justify its use. |
| 0 | Page 3 |



| Office Use Only |
|-----------------|
| Date Received: |
| Protocol Number |

☑ No – Skip to question 25 below

- 23. Who will have access to the identifiers and who will keep the link?
- 24. How will you limit access to the subject identifiers?
- 25. Describe the security plan for data including where it will be stored and how long, noting that you many not keep identifiable data indefinitely. All data obtained will be kept confidential in accordance with the provision of title 42 Code of Federal Regulations and HIPPA. All hard copy information will be kept in locked files, in locked rooms only accessible by Dr. Roh. All data collected during the study will be entered into an electronic data system by a unique ID code that will be assigned to each participant. Access to computer files will be only Dr. Roh. All data will be maintained in a computerized data system on a secured and firewall protected server. Hard copies of the focus group and interview transcripts, notes, and surveys will be kept in locked cabinets for 3 years in the USD Department of Social Work.

| Results from the study will be provided in the aggregate to avoid identification of a when there are not sufficient cases to assure confidentiality or when characteristic include any identifying information on participants and no participant-specific information. | s clearly identify a particular participant. No reports will |
|---|---|
| 26. Do you agree to keep a copy of the de-identified data for 3 years after the s ☐ Yes ☐ No Most exempt studies require a participant to be given a consent statement or a | • |
| most exempt studies require a participant to be given a consent statement of a | Cover letter. |
| <ul> <li>27. Check (✓) all that apply. Prepare and attach forms/scripts for review.</li> <li>□ Parental Consent (If the research is on a minor, parental conser sign the parental consent if it is written at a low literacy level.)</li> <li>☑ Informed Consent (Adults)</li> </ul> | nt is required. If minors are over 12 they can also |
| <ul> <li>☐ Assent Written (If child is ages 7-11 a written assent or verbal a</li> <li>☐ Assent-written within parental consent</li> <li>☐ Assent-verbal, script needed</li> </ul> | ssent is required. Verbal assent requires a script.) |
| <ul> <li>□ Consent Statement (This can only be used on adults when no id</li> <li>□ Cover Letter (This is similar to the consent statement but is in le</li> </ul> | |
| Templates can be found at <a href="http://www.usd.edu/research/irb-application-for">http://www.usd.edu/research/irb-application-for</a> regulatory compliance and avoid delays in processing this application. | rms. Please utilize the templates to ensure |
| | the consent?<br>Verbal/Handout (face to face<br>Verbal (telephone) |
| 29. Describe what will be said to the participant to introduce the research. If you must include a telephone script. You are invited to participate in a research stu evaluate the feasibility and effectiveness of the Mobile Web App Breast Cancer Schallored for Al women. In order to participate, you must be 40 or older Al women. The Please take time to read this flyer and ask questions before deciding whether to take the participant to introduce the research. If you must include a telephone script. You are invited to participate in a research students. | our study is a telephone survey or interview, you ady. The purpose of this study is to develop and creening (wMammogram) intervention that is culturally raking part in this research project is voluntary. |
| Section 4: Risks and Benefits | |
| 30. Are there any of the following risks associated with the research? Please on the control of | check all that apply.<br>□ Physical Risk<br>□ Psychological Risk<br>□ Social Risk |
| | Page 4 |



| Office Use Only |
|-----------------|
| Date Received: |
| Protocol Number |

| | ust send a copy of this section to the IRB office to complete your application. You | |
|---|---|---|
| | Signature Page | |
| 35. | 35. Does your study require HIPAA authorization or Waivers? □ N/A □ Full Waiver <a href="http://www.usd.edu/research/irb-general-forms">http://www.usd.edu/research/irb-general-forms</a> □ Partial Waiver <a href="http://www.usd.edu/research/irb-general-forms">http://www.usd.edu/research/irb-general-forms</a> □ Authorization Addendum (A study-specific Research Subjection (stand-alone) form must be attached) | rms |
| 34. | 34. Check PHI that you are collecting Names Email addresses Device identifiers Web universal resource Any unique identifying serial numbers Geographical subdivisions smaller than a State, including serial numbers than a State, including serial numbers than a State, including serial numbers of dates related to the individual, i.e. birthdate, and Health plan beneficiary numbers; account numbers; certifice Vehicle identifiers and serial numbers, including license plant | dmission date, discharge date, death.<br>cate/license numbers |
| | A authorizations or waivers may be appropriate if you are collecting F<br>cal center, doctor's office etc. | Protected Health Information (PHI) from a hospital, |
| 33. | <ul> <li>33. Have you notified all areas (personnel and facilities) that need to be portion in the properties of the pr</li></ul> | repared to assist you in your research? |
| | <ul><li>31. If you checked any boxes above, describe the nature of each risk and be present in the consent form. Click here to enter text.</li><li>32. What direct and societal benefits do you expect the subject(s) you enr benefit to the subjects, simply state that. There is no direct benefit to</li></ul> | roll to receive from this study? If there is no direct |
| | <ul> <li>☐ Use of private records including educational records or me</li> <li>☐ Collection of information that would be reportable to author subject prosecutable under the law (e.g. child abuse, alcohol a self or others.)</li> </ul> | rities or collection of information that might render the |

Dakota, Office of Human Subjects Protection, 414 E. Clark, Slagle Hall 107, Vermillion, SD 57069.

Title of Study: Intervention to Promote Breast Cancer Screening Among American Indian Women

Investigator(s) Name: Soonhee Roh, PhD

By signing below, I attest that the information provided in this form is correct. I agree to seek and obtain prior written approval from the IRB for any substantive modifications in the proposal, including changes in procedure, co-investigators, consent statements, survey/interview questions, etc. I will immediately report any unexpected or unanticipated problems or incidents that occur during the study. I will report in writing any significant findings which develop during the course of the study which may affect the risks and benefits to the participants. I will not begin my research until I have received approval from the IRB. I will abide by the IRB requests for to report on the status of the study. I will maintain the records and documents of this research. If there is a grant associated with this research, it completely reflects what is contained in this application. If the above conditions are not met, I understand that approval of this research could be suspended or terminated.



Office Use Only
Date Received:
Protocol Number

| Principal Investigator Signature: Soonhee Rah | 08/7/2019 |
|---|---|
| Thirty and the second s | Date |
| Student Investigator Signature: | |
| | Date |
| Honors Director and Department Chair or Dean Assurances: | |
| By signing below, I attest that I reviewed the above application and fir competencies and resources are adequate. | nd the research is scientifically and scholarly sound and that |
| Honors Director Signature: | |
| Signature | Date |
| By signing below, I attest that I reviewed the above application and fir competencies and resources are adequate. | nd the research is scientifically and scholarly sound and that |
| Department Chair or Dean Signature: | |
| Front Zoradil August 8, 2019, Signature Da | |
| Signature Da | lC |

### Submission Type: Modification Date: 2-4-2025

IRB #: 2019-053

Title: Exped-Intervention to Promote Breast Cancer Screening Among American Indian Women

Creation Date: 7-1-2021 Status: Review Complete

Principal Investigator: Soon Hee Roh

### Project Update/Amendment Form

### Select how your initial submission was made:

Cayuse

✓ Paper form or A-Tune

# Legacy Data: Amendment Form

| alla. | | |
|-------|-----|----|
| *req | uir | ed |

# 1. What are you revising?

Is the change significant?

3.

| | ✓ | Consent Form |
|----------|---|----------------------------------|
| | | Advertisements |
| | | Questionnaire/Survey |
| | | Adding a site or location |
| | | Investigator Brochure |
| | | Letter(s) of permission |
| | | IRB approvals other than USD IRB |
| | | Administrative letter |
| | | Closed to accrual |
| | | Other |
| 2. | С | hange of Personnel: |
| _ | | |
| | | Add Personnel |
| | | Remove Personnel |
| *require | d | |

| le | ease describe the change. |
|---|---|
| Υ | ade separate informed consent form both control and experimental group. |
| ۷I | nat is the reason for the change? |
| 0 | more effective intervention |
| ءاد | www.uld the proposed revision change the level of rick to the aubicate? |
| _ | w would the proposed revision change the level of risk to the subjects? |
| | Increase |
| | Decrease |
| | No change |

Yes

| * | | | | -1 |
|----|-----------------|-------|-----|----------|
| ** | $r \triangle c$ | 11 11 | ıre | $\alpha$ |

### 8. Are there changes needed to the consent form?

Attach a copy of the revised consent with the changes tracked or underlined and a clean copy for the IRB date-stamp at the bottom.

Do you have subjects enrolled with the previous consent?

Yes

✓ No

No

### 9. Attach all modified/updated documents:

✓ Informed Consent

Telephone scripts

Protocols from sponsors

Investigator brochure

Advertisements, flyers, posters

Surveys, questionnaires, interview questions

updated and original IRB application

CITI certificates

Final-0527-2021-Experimental Group Informed consent form.doc

Roh\_Consent\_Control Group by SHR-052621-Submit to JS.doc

#### \*required

### **Principal Investigator**

Name: Soon Hee Roh Organization: Social Work

Address: 1400 W 22nd Street SF HSC, Sioux Falls, SD 57105-1570

Phone: 605-357-1450

Email: soonhee.roh@usd.edu

#### \*required

### **Primary Contact**

Name: Serene Thin Elk Organization: Psychiatry

Address: , Vermillion, SD 57069-2390

Phone:

Email: serene.thinelk@gmail.com

### Co-Investigator(s)

Name: Yeon-Shim Lee

Organization: External IRB Study Address: , Vermillion, SD 57069-2390

Phone:

Email: YL375@sfsu.edu

Name: Shasheen Thin Elk

Organization: External IRB Study Address: , Vermillion, SD 57069-2390

Phone:

Email: SthinElk@yanktonsiouxtribe.net

# Student Investigator(s)

Name: Johanna Tietze

Organization: IRB Student Users

Address: , Vermillion, SD 57069-2390

Phone:

Email: Johanna.Tietze@coyotes.usd.edu

### **Study Documents**

 ${\color{blue} 2019.053-} Roh Lee\_Intervention to Promote... American Indian Women.pdf$ 

### Submission Type: Modification Date: 2-4-2025

IRB #: 2019-053

Title: Exped-Intervention to Promote Breast Cancer Screening Among American Indian Women

Creation Date: 10-1-2021 Status: Review Complete

Principal Investigator: Soon Hee Roh

### Project Update/Amendment Form

### Select how your initial submission was made:

Cayuse

✓ Paper form or A-Tune

# Legacy Data: Amendment Form

| alla. | |
|-------|-------|
| ~rec | uired |
| | 01100 |

# 1. What are you revising?

| ✓ | Consent Form |
|---|----------------------------------|
| ✓ | Advertisements |
| ✓ | Questionnaire/Survey |
| | Adding a site or location |
| | Investigator Brochure |
| | Letter(s) of permission |
| | IRB approvals other than USD IRB |
| | Administrative letter |
| | Closed to accrual |
| | Other |
| С | hange of Personnel: |
| | Add Personnel |
| | Remove Personnel |

\*required

2.

3. Is the change significant?

\*required

### Please describe the change.

There were minor grammatical changes made the consent statements and pre-test. There

4. were also changes to the participant payment information and include both informed consent forms and the updated flyers. Additionally, we changed our post-test based on our usability test and community advisory board members' suggestions and added sections VIII and IX and have a safety plan listed in the consent statements. We added an additional language as follow "If you may find some of the questions to be sensitive in nature or experience emotional discomfort, you can reach out to a licensed counselor at the Helpline Center (

1-800-273-8255)". This information will be included in the informed consent form.

\*required

### What is the reason for the change?

5.

Based on input and suggestions from our usability test and community advisory board members, we included additional questions that have been associated with cancer care and health behaviors.

\*required

6. How would the proposed revision change the level of risk to the subjects?

Increase

Decrease

| | d | |
|---|---|---|
| | Will th | nis have an impact on the study and/or participants? |
| | Yes | |
| • | ✓ No | |
| ec | | |
| | Are th | nere changes needed to the consent form? |
| | / Yes | <b>.</b> |
| • | <b>∕</b> Yes | |
| • | <b>√</b> Yes | Attach a copy of the revised consent with the changes tracked or underlined a clean copy for the IRB date-stamp at the bottom. |
| • | ✓ Yes | Attach a copy of the revised consent with the changes tracked or underlined |
| • | ✓ Yes | Attach a copy of the revised consent with the changes tracked or underlined |
| • | <b>√</b> Yes | Attach a copy of the revised consent with the changes tracked or underlined a clean copy for the IRB date-stamp at the bottom. Do you have subjects enrolled with the previous consent? |
| • | ✓ Yes | Attach a copy of the revised consent with the changes tracked or underlined a clean copy for the IRB date-stamp at the bottom. Do you have subjects enrolled with the previous consent? Yes |
| | ✓ Yes | Attach a copy of the revised consent with the changes tracked or underlined a clean copy for the IRB date-stamp at the bottom. Do you have subjects enrolled with the previous consent? |
| | ✓ Yes | Attach a copy of the revised consent with the changes tracked or underlined a clean copy for the IRB date-stamp at the bottom. Do you have subjects enrolled with the previous consent? Yes |
| | ✓ Yes | Attach a copy of the revised consent with the changes tracked or underlined a clean copy for the IRB date-stamp at the bottom. Do you have subjects enrolled with the previous consent? Yes |
| | _ | Attach a copy of the revised consent with the changes tracked or underlined a clean copy for the IRB date-stamp at the bottom. Do you have subjects enrolled with the previous consent? Yes |
| | _ | Attach a copy of the revised consent with the changes tracked or underlined a clean copy for the IRB date-stamp at the bottom. Do you have subjects enrolled with the previous consent? Yes |

✓ No change

Telephone scripts

Protocols from sponsors

Investigator brochure

- ✓ Advertisements, flyers, posters
- ✓ Surveys, questionnaires, interview questions updated and original IRB application

CITI certificates

2021---wMammogram flyer-submit -100121 for stamp .doc

Control Group Informed Consent Form-Clean version for stamp-100121.doc

Control Group Informed Consent Form-track change version-100121.doc

Control-Brochure-FINAL-9-30-21.pdf

Experiment GP-Informed Consent Form-Clean version for stamp-100121.doc

Experiment GP-Informed Consent Form-Track change version-100121.doc

Post-test Control Group-100121.doc

post-test-mobile web app -Experiment GP-100121.doc

Pre-test-all participants-100121.doc

USD IRB Amendment Application-100121.docx

#### \*required

### **Principal Investigator**

Name: Soon Hee Roh Organization: Social Work

Address: 1400 W 22nd Street SF HSC, Sioux Falls, SD 57105-1570

Phone: 605-357-1450

Email: soonhee.roh@usd.edu

#### \*required

### **Primary Contact**

Name: Serene Thin Elk Organization: Psychiatry

Address: , Vermillion, SD 57069-2390

Phone:

Email: serene.thinelk@gmail.com

### Co-Investigator(s)

Name: Yeon-Shim Lee

Organization: External IRB Study Address: , Vermillion, SD 57069-2390

Phone:

Email: YL375@sfsu.edu

Name: Shasheen Thin Elk

Organization: External IRB Study Address: , Vermillion, SD 57069-2390

Phone:

Email: SthinElk@yanktonsiouxtribe.net

# Student Investigator(s)

Name: Johanna Tietze

Organization: IRB Student Users

Address: , Vermillion, SD 57069-2390

Phone:

Email: Johanna.Tietze@coyotes.usd.edu

### **Study Documents**

 ${\color{blue} 2019.053-} Roh Lee\_Intervention to Promote... American Indian Women.pdf$ 

### Submission Type: Modification Date: 2-4-2025

IRB #: 2019-053

Title: Exped-Intervention to Promote Breast Cancer Screening Among American Indian Women

Creation Date: 5-2-2022 Status: Review Complete

Principal Investigator: Soon Hee Roh

### Project Update/Amendment Form

### Select how your initial submission was made:

Cayuse

✓ Paper form or A-Tune

# Legacy Data: Amendment Form

| alla. | | |
|-------|-----|----|
| *req | uir | ed |

# 1. What are you revising?

| | Consent Form |
|---|----------------------------------|
| ✓ | Advertisements |
| | Questionnaire/Survey |
| | Adding a site or location |
| | Investigator Brochure |
| | Letter(s) of permission |
| | IRB approvals other than USD IRB |
| | Administrative letter |
| | Closed to accrual |
| | Other |
| С | hange of Personnel: |

## Add Personnel

Remove Personnel

\*required

2.

3. Is the change significant?

| • | ✓ No |
|---|---|
| ec | d<br>d |
| | Please describe the change. |
| | We have 2 days of focus group meetings instead of one day meeting. |
| ec | 4 |
| | What is the reason for the change? |
| | Prospective focus group members request more time slots for their attendance. |
| ec | How would the proposed revision change the level of risk to the subjects? |
| | Tiow would the proposed revision change the level of fisk to the subjects: |
| | Increase |
| | Decrease |
| • | ✓ No change |
| | 4 |
| e | Will this have an impact on the study and/or participants? |

Yes

| * | rρ | ai | н | re | Ы |
|---|----|----|---|----|---|

### 8. Are there changes needed to the consent form?

Yes

✓ No

### Attach all modified/updated documents:

9.

Include the track changes version and a clean version in word format.

Informed Consent

Telephone scripts

Protocols from sponsors

Investigator brochure

✓ Advertisements, flyers, posters

Surveys, questionnaires, interview questions

updated and original IRB application

CITI certificates

Final-Follow-up focus group flyer-042722-request to Announcer.doc

Final-Follow-up focus group flyer-042722-request to Announcer.pdf

| Attach | other | approved | documents | associated | with this | modification. |
|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|

10.

(Only attach current approved versions)

#### \*required

### **Principal Investigator**

Name: Soon Hee Roh Organization: Social Work

Address: 1400 W 22nd Street SF HSC, Sioux Falls, SD 57105-1570

Phone: 605-357-1450

Email: soonhee.roh@usd.edu

#### \*required

### **Primary Contact**

Name: Serene Thin Elk Organization: Psychiatry

Address: , Vermillion, SD 57069-2390

Phone:

Email: serene.thinelk@gmail.com

### Co-Investigator(s)

Name: Yeon-Shim Lee

Organization: External IRB Study Address: , Vermillion, SD 57069-2390

Phone:

Email: YL375@sfsu.edu

Name: Shasheen Thin Elk

Organization: External IRB Study Address: , Vermillion, SD 57069-2390

Phone:

Email: SthinElk@yanktonsiouxtribe.net

# Student Investigator(s)

Name: Johanna Tietze

Organization: IRB Student Users

Address: , Vermillion, SD 57069-2390

Phone:

Email: Johanna.Tietze@coyotes.usd.edu

### **Study Documents**

 ${\color{blue} 2019.053-} Roh Lee\_Intervention to Promote... American Indian Women.pdf$ 

### Submission Type: Modification Date: 2-4-2025

IRB #: 2019-053

Title: Exped-Intervention to Promote Breast Cancer Screening Among American Indian Women

Creation Date: 7-1-2021 Status: Review Complete

Principal Investigator: Soon Hee Roh

### Project Update/Amendment Form

### Select how your initial submission was made:

Cayuse

✓ Paper form or A-Tune

# Legacy Data: Amendment Form

| alla. | | |
|-------|-----|----|
| *req | uir | ed |

# 1. What are you revising?

Is the change significant?

3.

| | ✓ | Consent Form |
|-----------|---|----------------------------------|
| | | Advertisements |
| | | Questionnaire/Survey |
| | | Adding a site or location |
| | | Investigator Brochure |
| | | Letter(s) of permission |
| | | IRB approvals other than USD IRB |
| | | Administrative letter |
| | | Closed to accrual |
| | | Other |
| 2. | С | hange of Personnel: |
| _ | | |
| | | Add Personnel |
| | | Remove Personnel |
| *required | | |

| lε | ease describe the change. |
|----|-------------------------------------------------------------------------|
| n | ade separate informed consent form both control and experimental group. |
| ۷ł | nat is the reason for the change? |
| or | more effective intervention |
| lo | w would the proposed revision change the level of risk to the subjects? |
| | ncrease |
| ľ | Decrease |
| ı | No change |

Yes

| * | | : | | -1 |
|----|-----------------|---|----|----------|
| ** | $r \triangle c$ | ш | re | $\alpha$ |

### 8. Are there changes needed to the consent form?

Attach a copy of the revised consent with the changes tracked or underlined and a clean copy for the IRB date-stamp at the bottom.

Do you have subjects enrolled with the previous consent?

Yes

✓ No

No

### 9. Attach all modified/updated documents:

✓ Informed Consent

Telephone scripts

Protocols from sponsors

Investigator brochure

Advertisements, flyers, posters

Surveys, questionnaires, interview questions

updated and original IRB application

CITI certificates

Final-0527-2021-Experimental Group Informed consent form.doc

Roh\_Consent\_Control Group by SHR-052621-Submit to JS.doc

#### \*required

### **Principal Investigator**

Name: Soon Hee Roh Organization: Social Work

Address: 1400 W 22nd Street SF HSC, Sioux Falls, SD 57105-1570

Phone: 605-357-1450

Email: soonhee.roh@usd.edu

#### \*required

### **Primary Contact**

Name: Serene Thin Elk Organization: Psychiatry

Address: , Vermillion, SD 57069-2390

Phone:

Email: serene.thinelk@gmail.com

### Co-Investigator(s)

Name: Yeon-Shim Lee

Organization: External IRB Study Address: , Vermillion, SD 57069-2390

Phone:

Email: YL375@sfsu.edu

Name: Shasheen Thin Elk

Organization: External IRB Study Address: , Vermillion, SD 57069-2390

Phone:

Email: SthinElk@yanktonsiouxtribe.net

# Student Investigator(s)

Name: Johanna Tietze

Organization: IRB Student Users

Address: , Vermillion, SD 57069-2390

Phone:

Email: Johanna.Tietze@coyotes.usd.edu

### **Study Documents**

 ${\color{blue} 2019.053-} Roh Lee\_Intervention to Promote... American Indian Women.pdf$ 

### Submission Type: Modification Date: 2-4-2025

IRB #: 2019-053

Title: Exped-Intervention to Promote Breast Cancer Screening Among American Indian Women

Creation Date: 10-1-2021 Status: Review Complete

Principal Investigator: Soon Hee Roh

### Project Update/Amendment Form

### Select how your initial submission was made:

Cayuse

✓ Paper form or A-Tune
# Legacy Data: Amendment Form

| alla. | |
|-------|-------|
| ~rec | uired |
| | 01100 |

# 1. What are you revising?

| ✓ | Consent Form |
|---|----------------------------------|
| ✓ | Advertisements |
| ✓ | Questionnaire/Survey |
| | Adding a site or location |
| | Investigator Brochure |
| | Letter(s) of permission |
| | IRB approvals other than USD IRB |
| | Administrative letter |
| | Closed to accrual |
| | Other |
| С | hange of Personnel: |
| | Add Personnel |
| | Remove Personnel |

\*required

2.

3. Is the change significant?

\*required

### Please describe the change.

There were minor grammatical changes made the consent statements and pre-test. There

4. were also changes to the participant payment information and include both informed consent forms and the updated flyers. Additionally, we changed our post-test based on our usability test and community advisory board members' suggestions and added sections VIII and IX and have a safety plan listed in the consent statements. We added an additional language as follow "If you may find some of the questions to be sensitive in nature or experience emotional discomfort, you can reach out to a licensed counselor at the Helpline Center (

1-800-273-8255)". This information will be included in the informed consent form.

\*required

### What is the reason for the change?

5.

Based on input and suggestions from our usability test and community advisory board members, we included additional questions that have been associated with cancer care and health behaviors.

\*required

6. How would the proposed revision change the level of risk to the subjects?

Increase

Decrease

| | ed | |
|---|---|---|
| | Will t | his have an impact on the study and/or participants? |
| | Ye | S. |
| | ✓ No | |
| | <b>∀</b> INU | |
| 1 | ed | |
| | Are t | here changes needed to the consent form? |
| | <b>√</b> Ye | S |
| | <b>√</b> Ye | |
| | <b>√</b> Ye | |
| | <b>√</b> Ye | Attach a copy of the revised consent with the changes tracked or underlined |
| | ✓ Ye | Attach a copy of the revised consent with the changes tracked or underlined |
| | ✓ Ye | Attach a copy of the revised consent with the changes tracked or underlined a clean copy for the IRB date-stamp at the bottom. |
| | ✓ Ye | Attach a copy of the revised consent with the changes tracked or underlined a clean copy for the IRB date-stamp at the bottom. Do you have subjects enrolled with the previous consent? Yes |
| | ✓ Ye | Attach a copy of the revised consent with the changes tracked or underlined a clean copy for the IRB date-stamp at the bottom. Do you have subjects enrolled with the previous consent? |
| | _ | Attach a copy of the revised consent with the changes tracked or underlined a clean copy for the IRB date-stamp at the bottom. Do you have subjects enrolled with the previous consent? Yes No |
| | ✓ Ye | Attach a copy of the revised consent with the changes tracked or underlined a clean copy for the IRB date-stamp at the bottom. Do you have subjects enrolled with the previous consent? Yes No |
| | _ | Attach a copy of the revised consent with the changes tracked or underlined a clean copy for the IRB date-stamp at the bottom. Do you have subjects enrolled with the previous consent? Yes No |
| | _ | Attach a copy of the revised consent with the changes tracked or underlined a clean copy for the IRB date-stamp at the bottom. Do you have subjects enrolled with the previous consent? Yes No |

✓ No change

Telephone scripts

Protocols from sponsors

Investigator brochure

- ✓ Advertisements, flyers, posters
- ✓ Surveys, questionnaires, interview questions updated and original IRB application

CITI certificates

2021---wMammogram flyer-submit -100121 for stamp .doc

Control Group Informed Consent Form-Clean version for stamp-100121.doc

Control Group Informed Consent Form-track change version-100121.doc

Control-Brochure-FINAL-9-30-21.pdf

Experiment GP-Informed Consent Form-Clean version for stamp-100121.doc

Experiment GP-Informed Consent Form-Track change version-100121.doc

Post-test Control Group-100121.doc

post-test-mobile web app -Experiment GP-100121.doc

Pre-test-all participants-100121.doc

USD IRB Amendment Application-100121.docx

### \*required

## **Principal Investigator**

Name: Soon Hee Roh Organization: Social Work

Address: 1400 W 22nd Street SF HSC, Sioux Falls, SD 57105-1570

Phone: 605-357-1450

Email: soonhee.roh@usd.edu

#### \*required

### **Primary Contact**

Name: Serene Thin Elk Organization: Psychiatry

Address: , Vermillion, SD 57069-2390

Phone:

Email: serene.thinelk@gmail.com

### Co-Investigator(s)

Name: Yeon-Shim Lee

Organization: External IRB Study Address: , Vermillion, SD 57069-2390

Phone:

Email: YL375@sfsu.edu

Name: Shasheen Thin Elk

Organization: External IRB Study Address: , Vermillion, SD 57069-2390

Phone:

Email: SthinElk@yanktonsiouxtribe.net

# Student Investigator(s)

Name: Johanna Tietze

Organization: IRB Student Users

Address: , Vermillion, SD 57069-2390

Phone:

Email: Johanna.Tietze@coyotes.usd.edu

### **Study Documents**

 ${\color{blue} 2019.053-} Roh Lee\_Intervention to Promote... American Indian Women.pdf$ 

### Submission Type: Modification Date: 2-4-2025

IRB #: 2019-053

Title: Exped-Intervention to Promote Breast Cancer Screening Among American Indian Women

Creation Date: 5-2-2022 Status: Review Complete

Principal Investigator: Soon Hee Roh

### Project Update/Amendment Form

## Select how your initial submission was made:

Cayuse

✓ Paper form or A-Tune

# Legacy Data: Amendment Form

| alla. | | |
|-------|------|---|
| *req | uire | Ν |

# 1. What are you revising?

| | Consent Form |
|---|----------------------------------|
| ✓ | Advertisements |
| | Questionnaire/Survey |
| | Adding a site or location |
| | Investigator Brochure |
| | Letter(s) of permission |
| | IRB approvals other than USD IRB |
| | Administrative letter |
| | Closed to accrual |
| | Other |
| С | hange of Personnel: |

## Add Personnel

Remove Personnel

\*required

2.

3. Is the change significant?

| Pl | ease describe the change. |
|---|---|
| W | e have 2 days of focus group meetings instead of one day meeting. |
| W | hat is the reason for the change? |
| Pr | ospective focus group members request more time slots for their attendance. |
| d | |
| Н | ow would the proposed revision change the level of risk to the subjects? |
| | Increase |
| | Decrease |
| / | No change |

Yes

| * | rρ | ai | н | re | Ы |
|---|----|----|---|----|---|

### 8. Are there changes needed to the consent form?

Yes

✓ No

### Attach all modified/updated documents:

9.

Include the track changes version and a clean version in word format.

Informed Consent

Telephone scripts

Protocols from sponsors

Investigator brochure

✓ Advertisements, flyers, posters

Surveys, questionnaires, interview questions

updated and original IRB application

CITI certificates

Final-Follow-up focus group flyer-042722-request to Announcer.doc

Final-Follow-up focus group flyer-042722-request to Announcer.pdf

| Attach | other | approved | documents | associated | with this | modification. |
|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|

10.

(Only attach current approved versions)

### \*required

## **Principal Investigator**

Name: Soon Hee Roh Organization: Social Work

Address: 1400 W 22nd Street SF HSC, Sioux Falls, SD 57105-1570

Phone: 605-357-1450

Email: soonhee.roh@usd.edu

#### \*required

### **Primary Contact**

Name: Serene Thin Elk Organization: Psychiatry

Address: , Vermillion, SD 57069-2390

Phone:

Email: serene.thinelk@gmail.com

### Co-Investigator(s)

Name: Yeon-Shim Lee

Organization: External IRB Study Address: , Vermillion, SD 57069-2390

Phone:

Email: YL375@sfsu.edu

Name: Shasheen Thin Elk

Organization: External IRB Study Address: , Vermillion, SD 57069-2390

Phone:

Email: SthinElk@yanktonsiouxtribe.net

# Student Investigator(s)

Name: Johanna Tietze

Organization: IRB Student Users

Address: , Vermillion, SD 57069-2390

Phone:

Email: Johanna.Tietze@coyotes.usd.edu

### **Study Documents**

 ${\color{blue} 2019.053-} Roh Lee\_Intervention to Promote... American Indian Women.pdf$